CLINICAL TRIAL: NCT04348799
Title: Thrombocytopoiesis and Platelet Homeostasis in Infants With Bronchoplumonary Dysplasia
Acronym: BPD
Status: Completed | Type: Observational
Sponsor: yangjie (Other)
Responsible Party: Sponsor-Investigator, yangjie, Director of Dept of Neonatology, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Other Study IDs: Guangdong W C H
Record Dates: First submitted 2020-03-15; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Bronchopulmonary Dysplasia; Thrombocytopenia; Preterm Infant
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Thrombocytopenia; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral arterial blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPD group: premature infants diagnosed with BPD after postnatal day 28
  Interventions: Other: BPD
- control group: premature infants without BPD after postnatal day 28

INTERVENTIONS:
Other: BPD — It is a observation research.we didn't intervene anything.
  Groups: BPD group

SUMMARY:
To investigate the relationship between bronchopulmonary dysplasia and thrombocytopenia.

DETAILED DESCRIPTION:
A prosepective case-control study ,the case were matched with 1:1according to gestational age,birth weight and admission diagnosis and divided into two groups according to the consensus definition of National Institute of Child Health and Human Development (NICHD). Platelet count, circulating megakaryocyte count, platelet activating markers (CD62P and CD63), thrombopoietin were recorded and compared in two groups, then, serial thrombopoietin levels and concomitant platelet counts were measured in infants with BPD.

ELIGIBILITY:
Inclusion Criteria:

1. presence of clinical and radiologic signs of BPD, according to conventional criteria (Greenough, 1992);
2. presence of peripheral arterial catheter;
3. gestation <32 weeks;
4. birth weight <1.5 kg;
5. requiring mechanical ventilation for the treatment of respiratory distress syndrome for at least 3 days during the first weeks of life;
6. ventilator and/or oxygen dependent at time of enrolment;

Exclusion Criteria:

1. congenital abnormalities;
2. infection (bacteria infection confirmed by positive blood culture or viral infection confirmed by serological test or viral culture)
3. evidence of complications of perinatal asphyxia including an apgar score <3 at one or five minute after birth, evidence of hypoxic-ischemic encephalopathy, acute tubular necrosis, or transient myocardial ischemia;
4. identifiable hematologic disease;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Bronchopulmonary dysplasia (BPD) is one of the common complications in neonatal intensive care units (NICU), mainly occurs in premature infants and is considered to be the main cause of premature death
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Platelet counts and Circulating MK counts | up to 4 weeks
  Platelet counts and Circulating MK counts

SECONDARY OUTCOMES:
CD62P and CD63 expression | up to 4 weeks
  CD62P and CD63 expression
TPO | up to 4 weeks
  Plasma TPO concentration
TPO and platelet | up to 6 weeks
  the relationship betweenTPO concentration and Platelet counts in BPD with thrombocytopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China